CLINICAL TRIAL: NCT02309294
Title: 14-Day Cumulative Irritation Patch Test in Subjects With Normal Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ST-7553
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Cumulative Irritation
Keywords: Patch Test

ARMS (1):
- Healthy Subject (Experimental): Occlusive patches applied each day for 14 days for each intervention (Experimental: Novel lubricant Miami w/ fragrance, Experimental: Novel lubricant Miami no fragrance, KY Liquid lubricant, Astroglide Gel lubricant, Wet Platinum lubricant).
  Interventions: Device: Novel lubricant Miami w/ fragrance; Device: Novel lubricant Miami no fragrance; Device: KY Liquid lubricant; Device: Astroglide Gel lubricant; Device: Wet Platinum lubricant

INTERVENTIONS:
Device: Novel lubricant Miami w/ fragrance — 0.2 ml aliquot on occlusive patch
Device: Novel lubricant Miami no fragrance — 0.2 ml aliquot on occlusive patch
Device: KY Liquid lubricant — 0.2 ml aliquot on occlusive patch
Device: Astroglide Gel lubricant — 0.2 ml aliquot on occlusive patch
Device: Wet Platinum lubricant — 0.2 ml aliquot on occlusive patch

SUMMARY:
The objective of this study is to determine the ability of the study material to cause irritation to the skin of humans under controlled patch test conditions. Substances that come into contact with human skin need to be evaluated for their propensity to irritate and/or sensitize. This testing is a modified primary irritancy patch test that can detect weak irritants that require multiple applications to cause a skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* Are a male or female, 18 years of age or older, in general good health;
* Have normal skin;
* Are free of any systemic or dermatologic disorder which, in the opinion of the investigative personnel, will interfere with the study results or increase the risk of adverse events;
* Are of any skin type or race providing the skin pigmentation will allow discernment of erythema;
* Complete a medical screening procedure; and
* Read, understand, and sign an informed consent.

Exclusion Criteria:

* Have any visible skin disease at the study site which, in the opinion of the investigative personnel, will interfere with the evaluation;
* Are receiving systematic or topical drugs or medication which, in the opinion of the investigative personnel, will interfere with the study results;
* Have psoriasis and/or active atopic dermatitis/eczema; and/or
* Have a known sensitivity to cosmetics, skin care products, or topical drugs as related to the material being evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Subject
Started | 43
Completed | 41
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 41
Age, Customized [Number; unit: participants]
  20-72 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Showed no Significant Irritation
Description: Score of less than or equal to 1.2 on the Cumulative Irritation Test scale (0-5).
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 41
participants | 0

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place